CLINICAL TRIAL: NCT05359341
Title: Comparative Study of DPP-4 Inhibitors and SGLT-2 Inhibitors in Egyptian Diabetic Patients
Brief Title: Which is Better to Start With DPP-4 Inhibitors or SGLT-2 Inhibitors in Egyptian Diabetic Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadat City University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Haitham Galal, Teaching assistant (MSC) in Clinical Pharmacy Department, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/2020
Record Dates: First submitted 2022-04-05; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; empagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sitagliptin 50 mg twice daily (Active Comparator): sitagliptin 50 mg is added for 12 weeks to T2DM not controlled with diet, exercise and metformin with or without other oral antidiabetic drugs.
  Interventions: Drug: Sitagliptin 50 mg
- Empagliflozin 12.5 twice daily (Active Comparator): Empagliflozin 12.5 mg is added for 12 weeks to T2DM not controlled with diet, exercise and metformin with or without other oral antidiabetic drugs.
  Interventions: Drug: Empagliflozin 12.5 MG
- Sitagliptin 50 mg + empagliflozin 12.5 mg (Active Comparator): empagliflozin 12.5 mg is added to the patients with HbA1c 7-10 % of sitagliptin 50 mg group for another 12 weeks.
  Interventions: Drug: Sitagliptin 50 mg + Empagliflozin 12.5 MG
- Empagliflozin 12.5 + sitagliptin 50mg (Active Comparator): sitagliptin 50 mg is added to the patients with HbA1c 7-10 % of empagliflozin 12.5 mg group for another 12 weeks.
  Interventions: Drug: Empagliflozin 12.5 MG + Sitagliptin 50 mg

INTERVENTIONS:
Drug: Sitagliptin 50 mg — Adding on sitagliptin to uncontrolled T2D Egyptian patients who are not controlled with diet, exercise and metformin with or without other OADs for 12 weeks.
  Other Names: DPP4 inhibitor
  Arms: Sitagliptin 50 mg twice daily
Drug: Empagliflozin 12.5 MG — Adding on empagliflozin to uncontrolled T2D Egyptian patients who are not controlled with diet, exercise and metformin with or without other OADs for 12 weeks.
  Other Names: SGLT2 inhibitor
  Arms: Empagliflozin 12.5 twice daily
Drug: Sitagliptin 50 mg + Empagliflozin 12.5 MG — Adding on another 12 weeks of therapy of empagliflozin to sitagliptin 50mg group not well controlled (HbA1c 7-10%)
  Other Names: DPP4 inhibitor + SGLT2 inhibitor
  Arms: Sitagliptin 50 mg + empagliflozin 12.5 mg
Drug: Empagliflozin 12.5 MG + Sitagliptin 50 mg — Adding on another 12 weeks of therapy of sitagliptin 50mg to empagliflozin group not well controlled (HbA1c 7-10%)
  Other Names: SGLT2 inhibitor + DPP4 inhibitor
  Arms: Empagliflozin 12.5 + sitagliptin 50mg

SUMMARY:
Our trial goal is to determine the efficacy and safety of sitagliptin in comparison with empagliflozin in type 2 diabetic Egyptian patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 male/female diabetic patients
* Age 20-70 years
* A1C less than 10.5%

Exclusion Criteria:

* Type 1 diabetes; HbA1c > 10.5%
* Pregnancy
* Chronic liver disease
* Elevated (more than twofold the upper limit of normal) ALT, AST and CPK.
* High bilirubin
* Albumin < 3.5 g/dl
* INR >1-2 Diabetic ketoacidosis
* Urinary tract infection (UTI)
* Pancreatitis < 6 months prior to enrolment
* Renal impairment (creatinine clearance ≤50 ml/min)
* Treatment with anti-obesity drugs or glucagon-like peptide-1 receptor agonists (GLP-1RAs) 3 months prior to enrolment
* Non-compliance with follow-up visits.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Proportion of cured patients in the sitagliptin group versus the proportion of cured patients in the empagliflozin group | After completion of the study (One year anticipated)
  The primary efficacy endpoint will be evaluated as clinical cure after 12 weeks of addition of sitagliptin or empagliflozin to metformin and after 12 weeks after adding empaglifozin to sitagliptin group and vise versa.
  Clinical cure defined by A1C controlled (less than 7%), decrease in fasting and postprandial plasma glucose (mg/dl).

SECONDARY OUTCOMES:
The decrease in the body weight in patients in sitagliptin group versus empagliflozin group | After completion of the study (One year anticipated)
  The decreased in body weight (Kg) from the baseline measures after therapy.
The decrease in blood pressure in patients in sitagliptin group versus empagliflozin group | After completion of the study (One year anticipated)
  decrease in blood pressure is defined as the decrease in SBP and/or DBP (mmHg) from the baseline measures after completing therapy
The change in lipid profile in patients in sitagliptin group versus empagliflozin group | After completion of the study (One year anticipated)
  Change in lipid profile including decreasing in the following measures from the baseline measures after therapy is completed: low density lipoprotein (mg/dl), total cholesterol (mg/dl), triglyceride (mg/dl) and high density lipoprotein (mg/dl).

OTHER OUTCOMES:
Percentage of adverse effects appeared in patients in sitagliptin group versus percentage of adverse effects appear in patients in the empagliflozin group. | After completion of the study (One year anticipated)
  AEs (n%) included all events with an onset after the first dose of open label emoagliflozin or sitagliptin and up to 7 days after the last dose of study drug. AEs of special interest included hypoglycaemia, genitourinary infections, hypersensitivity reactions, diabetic ketoacidosis, acute pancreatitis, hypotension, and dehydration. Confirmed hypoglycemic AEs were defined as events with a plasma glucose concentration of ≤ 3.9 mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sadat City, El Sadat, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol